CLINICAL TRIAL: NCT06730438
Title: Transcranial Pulse Stimulation: a Potential New Treatment for Chronic Disorders of Consciousness/Cognition Due to Vegetative/Minimally Conscious States and Early Dementia
Brief Title: Transcranial Pulse Stimulation. a Potential Treatment for Early Dementia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Francesca Pistoia (Other)
Responsible Party: Sponsor-Investigator, Francesca Pistoia, Associate Professor of Neurology, ASL 1 Avezzano Sulmona L'Aquila
Organization: ASL 1 Avezzano Sulmona L'Aquila (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PNRR-MCNT2-2023-12377235; PNRR-MCNT2-2023-12377235 (Other Grant/Funding Number: Ministry of Health (Italy))
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's disease; Transcranial Pulse Stimulation; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Double Blind Sham-Controlled Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transcranial pulse stimulation (Experimental): Patients belonging to this group will receive real transcranial pulse stimulation over a 4-weeks period, once a day for five days a week.
  Interventions: Device: Transcranial Pulse Stimulation
- Sham stimulation Group (Sham Comparator): Patients belonging to this group will receive sham transcranial pulse stimualtion over a 4-weeks period, once a day for five days a week.
  Interventions: Device: Transcranial Pulse Stimulation

INTERVENTIONS:
Device: Transcranial Pulse Stimulation — Patients will receive TPS once a day for five days a week, each session will be separated from the previous one by 24h. Each stimulation and assessment session will be performed at the same hour of the day, in the morning preferably, to maximize the probability of observing responses to stimuli. Patients will be managed in a quiete room with stable light and temperature.

SUMMARY:
Alzheimer's Disease (AD) is characterized by the absence of treatments to slow, stop, or reverse its course, with patients finally losing cognitive functions, skills and independence. It is a chronic degenerative disease with high social and medical burden worldwide: AD ranked third among neurological disorders in terms of disability-adjusted life years (DALY) rates.

The primary aim of the research protocol is to improve care for patients with AD, by implementing, with an innovative method, the currently available repertoire of neuromodulation techniques. For this aim, we will investigate whether Transcranial Pulse Stimulation (TPS) may induce cognitive improvement in patients with an early stage of dementia.

DETAILED DESCRIPTION:
Aims of the project: The primary aim of our research protocol is to improve care for patients with AD by investigating whether Transcranial Pulse Stimulation (TPS) may induce cognitive improvement in patients with an early stage of dementia. Additional aims will include the investigation of the neurophysiological profile of patients and the search for a correlation between neuropsychological and neurophysiological data with the serum levels of brain-derived neurotrophic factor (BDNF) and of vascular endothelial growth factor (VEGF).

Materials and Methods: Following a rigorous selection, included patients will be treated through a real/sham structured TPS protocol and followed-up with respect to cognitive improvement, by comparing baseline and follow-up clinical scores. A Double Blind Sham-Controlled Study will be performed: patients will be assigned randomly to receive TPS or sham TPS for 4 weeks in a parallel groups, double-blind study. Patients will receive ether TPS or sham treatment once a day for five days a week for the whole period and will be assessed according to the following schedule: baseline (t0); at two weeks following the start of TPS (t1); at 1 month following the start of TPS (t2); at 2 months following the start of TPS (t3); at 6 months following the start of TPS (t4). Electroencephalography (EEG) and Somatory Evoked Potentials (SEP) will be contextually recorded in all patients, to compare neurophysiological data of patients treated with real TPS and sham stimulation. Moreover, a serum sample will be collected from patients at baseline, at the end of the stimulation period and at the 6-month follow-up, to compare preprocedural and postprocedural levels of serum BDNF and VEGF.

ELIGIBILITY:
Inclusion Criteria:

* age>18 years
* diagnosis of early dementia according to current international guidelines
* disease duration of at least 12 months
* consent to participate in the study.

Exclusion Criteria:

* medical instability interfering with standard neurological assessment
* any contraindication to preliminary MRI for MR-based real-time neuronavigation
* comorbidities which may interfere with cognitive status
* any contraindication to Transcranial Pulse Stimulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Cognitive improvement | Two weeks following the start of TPS (t1); at 1 month following the start of TPS (t2); at 2 months following the start of TPS (t3); 6 months following the start of TPS (t4).
  Cognitive improvement as evaluated by means of the ADAS-Cog, scores range from 0, that means the absence of cognitive dysfunctions, to a maximum of 70, that indicates a serious deficit in all tests.

CONTACTS AND LOCATIONS:
Locations (1):
- San Salvatore Hospital, L’Aquila, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Matt E, Kaindl L, Tenk S, Egger A, Kolarova T, Karahasanovic N, Amini A, Arslan A, Saricicek K, Weber A, Beisteiner R. First evidence of long-term effects of transcranial pulse stimulation (TPS) on the human brain. J Transl Med. 2022 Jan 15;20(1):26. doi: 10.1186/s12967-021-03222-5. PMID 35033118
- [Background] Beisteiner R, Matt E, Fan C, Baldysiak H, Schonfeld M, Philippi Novak T, Amini A, Aslan T, Reinecke R, Lehrner J, Weber A, Reime U, Goldenstedt C, Marlinghaus E, Hallett M, Lohse-Busch H. Transcranial Pulse Stimulation with Ultrasound in Alzheimer's Disease-A New Navigated Focal Brain Therapy. Adv Sci (Weinh). 2019 Dec 23;7(3):1902583. doi: 10.1002/advs.201902583. eCollection 2020 Feb. PMID 32042569